CLINICAL TRIAL: NCT07028567
Title: Comparative Study of Subcision Followed by Diluted Calcium Hydroxylapatite Injection Versus Subcision Followed by Painting CROSS TCA Technique for the Treatment of Atrophic Acne Scars
Brief Title: Subcision Followed by Diluted Calcium Hydroxylapatite Injection Versus Subcision Followed by Painting CROSS TCA Technique for the Treatment of Atrophic Acne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Riham Mohamed ElSayed ElSetiha, Resident of Dermatology and Venereology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36195/12/22
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Subcision; Calcium Hydroxylapatite; Trichloroacetic Acid; Atrophic Acne Scar

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients with atrophic acne scars.
  Interventions: Drug: Calcium hydroxylapatite filler; Drug: Painting chemical reconstruction of skin scars trichloroacetic acid technique

INTERVENTIONS:
Drug: Calcium hydroxylapatite filler — Patients received calcium hydroxylapatite filler (CaHA) (Radiesse®).
Drug: Painting chemical reconstruction of skin scars trichloroacetic acid technique — Patients received painting chemical reconstruction of skin scars (CROSS) trichloroacetic acid (TCA) technique.

SUMMARY:
This study aimed to compare the safety and efficacy of subcision followed by diluted calcium hydroxyapatite injection versus subcision followed by the painting original chemical reconstruction of skin scars (CROSS) technique using trichloroacetic acid (TCA) for the treatment of atrophic acne scars.

DETAILED DESCRIPTION:
Atrophic scars present as depressions secondary to fibrous contractions. Subcision is a technique in which a needle is inserted under the acne scar to sever the fibrous tissue (tethers) that bind down the scar. This releases the fibrous tissue.

The original chemical reconstruction of skin scars (CROSS) technique using trichloroacetic acid (TCA) entails focal application of highly concentrated TCA (70% to 100%) with firm pressure applied to the entire atrophic area using a sharpened wooden applicator until frosting occurs.

Fillers containing hyaluronic acid, calcium hydroxyapatite, and poly-L-lactic acid are increasingly used to correct atrophic acne scarring as they augment soft tissue in variable degree and are most effective in soft rolling or boxcar scars.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 50 years.
* Both sexes.
* Patients with atrophic acne scars.

Exclusion Criteria:

* Patients with Fitzpatrick skin phototypes V and VI.
* Receiving systemic isotretinoin medication at the time of the study.
* Active bacterial, viral or fungal infections in the treatment area.
* Hypertrophic scarring or keloidal tendency.
* Photosensitivity or photodermatitis.
* Unrealistic expectation, bleeding, coagulation disorders, and any other related skin disease.
* Pregnant or lactating females.
* Chronic debilitating diseases such as diabetes mellitus, cardiovascular diseases, renal failure, hepatic diseases, chronic respiratory diseases or any endocrine diseases.
* History of immunosuppressive drug intake or chemotherapy within 6 months before treatment.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | One week
  Patient satisfaction was assessed at the final follow-up visit using a 5-point Likert-type scale, comparing outcomes to the pre-treatment condition. The scale ranged from 1 (highly dissatisfied), 2 (slightly dissatisfied), 3 (neither satisfied nor dissatisfied), 4 (satisfied), to 5 (highly satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.